CLINICAL TRIAL: NCT00756431
Title: Prospective Randomized Double Blinded Clinical Evaluation on HA Coated Dynamic Hip Screws for Trochanteric Femoral Fractures
Brief Title: Clinical Evaluation on HA Coated Dynamic Hip Screws for Trochanteric Femoral Fractures
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No data so far
Sponsor: Zimmer Biomet (Industry)
Collaborators: Hvidovre University Hospital (Other); Biomet U.K. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BMET UK 06
Record Dates: First submitted 2008-09-19; First posted 2008-09-22 (Estimated); Last update posted 2017-06-19 (Actual); Status verified 2017-06

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Screw without HA Coating (Hiploc) (Active Comparator)
  Interventions: Device: Hip Fracture reduction Screw without HA Coating (Hiploc)
- Screw with HA Coating (Hiploc) (Experimental)
  Interventions: Device: Hip Fracture reduction Screw with HA Coating (Hiploc)

INTERVENTIONS:
Device: Hip Fracture reduction Screw without HA Coating (Hiploc) — Hip Fracture reduction Screw without HA Coating (Hiploc)
  Other Names: Hiploc
  Arms: Screw without HA Coating (Hiploc)
Device: Hip Fracture reduction Screw with HA Coating (Hiploc) — Hip Fracture reduction Screw with HA Coating (Hiploc)
  Other Names: Hiploc
  Arms: Screw with HA Coating (Hiploc)

SUMMARY:
Evaluated whether HA coated dynamic hip screws can improve the surgical results in trochanteric femoral fractures

DETAILED DESCRIPTION:
Randomised study to determine the effect of HA coating on the stability of lag screws used to reduce femoral neck fractures. Stability of the screw will be determined by RSA measurements. The effect of the HA coating on bone remodeling will be determined by DEXA measurements

ELIGIBILITY:
Inclusion Criteria:

* Patients with trochanteric femoral fractures

Exclusion Criteria:

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2004-01; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Harris Hip Score | 3months, 6 months

SECONDARY OUTCOMES:
DEXA | 3months, 6 months
RSA | 3months,6 months
Complications | Anytime

CONTACTS AND LOCATIONS:
Overall Officials: Hendrik Palm, MD, Principal Investigator — Hvidovre Univ. Hospital